CLINICAL TRIAL: NCT00785330
Title: Open, Multicentral, Randomised Phase II Study of Allogene Stem Cell Transplantation After Pretreatment With Fludarabin, Busulfan, Cyclophospahmid and GVHD-prophylaxis With or Without Rituximab in Patients With Recidivation of High Grade Non-hodgkin's Lymphoma in Special Risk Situation in the Age of 18 - 65
Brief Title: Allo-hNHL (FluBuCy)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut fuer anwendungsorientierte Forschung und klinische Studien GmbH (Other)
Collaborators: University Hospital Goettingen (Other); German High-Grade Non-Hodgkin's Lymphoma Study Group (Other)
Responsible Party: Prof. Dr. med. Glass, University Hospital Goettingen, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSHNHL 2004-R3
Record Dates: First submitted 2005-09-13; First posted 2008-11-05 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: rituximab; Non-Hodgkin's lymphoma; diffuse large B cell lymphoma; peripheral t cell lymphoma; graft-versus-host disease; graft-versus-lymphoma effect; allogeneic haematopoietic stem cell transplantation; relapsed or primary progressive aggressive Non-Hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, T-Cell, Peripheral; Graft vs Host Disease; Recurrence | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Other): Patients receiving no rituximab as GVHD prophylaxis after allogeneic SZT and only standard GVHD prophylaxis (tacrolimus with aimed serum level of 10 ng / ml and mycophenolat mofetil 2 x 1 g p.o. day 1 to 28 after allogeneic SZT
  Interventions: Drug: standard GVHD prophylaxis
- B (Experimental): rituximab in addition to standard GVHD prophylaxis
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: standard GVHD prophylaxis — Application of tacrolimus from day -1 with a goal of tacrolimus serum concentration of 10 ng / ml Aplication of mycophenolat mofetil from day +1 to day +28 in a dose of 2 x 1g per day
  Arms: A
Drug: rituximab — Patients receiving 375 mg/ m2 of rituximab at weeks 3, 4, 5, 6, 25, 26, 27, 28 after allogeneic stem cell transplantation in addition to standard GVHD prophylaxis (tacrolimus with aimed serum level of 10 ng / ml and mycophenolat mofetil 2 x 1 g p.o. day 1 to 28 after allogeneic SZT
  Arms: B

SUMMARY:
DSHNHL R3 is a randomized clinical phase II study. The main objective is to estimate the efficacy of rituximab as a prophylactic medication for prevention of graft-versus-host-disease after allogeneic peripheral stem cell transplantation in patients with a high risk relapse of aggressive B-cell Non-Hodgkin's lymphoma. The most important secondary objective is to estimate the efficacy of allogeneic stem cell transplantation in this clinical situation.

DETAILED DESCRIPTION:
Patients in the age of 18 to 65 years with a high- risk relapse of a histology proven aggressive Non-Hodgkin's-lymphoma are eligible for the trial. Aggressive Non-Hodgkin's lymphoma within this study is defined as:

B-NHL:

follicular lymphoma grade III° lymphoblastic (precursor) lymphoma diffuse large cell cell lymphoma any subtype and variant including primary mediastinal lymphoma mantle cell lymphoma, blastic variant

T-NHL:

precursor T cell lymphoma peripheral T cell lymphoma, any subtype and variant angioimmunoblastic lymphoma anaplastic large cell lymphoma, any subtype NK / T cell lymphoma High risk relapsed or progressive disease is defined as (a) primary progressive disease, (b) early relapse after less than 12 month of remission duration and at least one risk factor according to the international prognostic index (IPI), (c) relapse or progression after high dose chemotherapy and autologous transplantation, (d) relapse or progression and lack of an autologous stem cell product.

Patients with this type of progression / relapse should receive rituximab plus ifosfamide/carboplatin/etoposide (R-ICE) or rituximab plus dexamethasone/high dose ARA-C/cisplatinum as salvage therapy (recommendation, not part of study medication). In patients biwth T cell lymphoma rituximab may be replaced by alemtuzumab. If at least stable disease is achieved, patients can be definitely included.

With inclusion, patients were randomized to receive either 375 mg/ m2 of rituximab at weeks 3, 4, 5, 6, 25, 26, 27, 28 after allogeneic stem cell transplantation or no additional medication.

Conditioning for transplantation consisted of Fludarabine 125 mg/m2, Busulfan 12 mg/kg and cyclophosphamide 120 mg/kg.

Short-term (day 1 to day 28) mycophenolat mofetil and tacrolimus are used as basis GVHD prophylaxis in all patients. Anti-thymocyte globulin can be used due to the centres decision in patients with unrelated donors

ELIGIBILITY:
Inclusion Criteria:

* histology proven aggressive non Hodgkin's lymphoma and
* primary progressive disease or
* early relapse after less than 12 month of remission duration and at least one risk factor according to the international prognostic index (IPI or
* relapse or progression after high dose chemotherapy and autologous transplantation or
* relapse or progression and lack of an autologous stem cell product.

Exclusion Criteria:

* severe comorbidity or impaired organ function
* hypersensitivity to used drugs
* HIV positivity
* active hepatitis
* other active malignant disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2004-04; Primary Completion 2009-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The specific measure that will be used to determine the effect of the intervention(s) or, for observational studies, related to core objectives of the study and receiving the most emphasis in assessment. (a) rate of acute GVHD grade II-IV after one year | One year after allogeneic stem cell transplantation

SECONDARY OUTCOMES:
progression free survival, progression rate, non-relapse mortality, rate of grade 3-4 infectious adverse event, chronic GVHD | one and three years after allogeneic SZT

CONTACTS AND LOCATIONS:
Overall Officials: Bertram Glass, Prof. MD., Study Director — Asklepios Klinik St. Georg
Locations (6):
- Germany (6):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Würtenberg
  - Universitätsklinikum Marburg, Marburg, Hesse
  - Universitätsklinikum und Poliklinik, Homburg, Saarland
  - University Hospital Goettingen, Göttingen
  - Asklepios Klinik St. Georg, Hamburg
  - KMT-Zentrum Medizinische Klinik A, Münster

REFERENCES:
- [Derived] Glass B, Hasenkamp J, Wulf G, Dreger P, Pfreundschuh M, Gramatzki M, Silling G, Wilhelm C, Zeis M, Gorlitz A, Pfeiffer S, Hilgers R, Truemper L, Schmitz N; German High-Grade Lymphoma Study Group. Rituximab after lymphoma-directed conditioning and allogeneic stem-cell transplantation for relapsed and refractory aggressive non-Hodgkin lymphoma (DSHNHL R3): an open-label, randomised, phase 2 trial. Lancet Oncol. 2014 Jun;15(7):757-66. doi: 10.1016/S1470-2045(14)70161-5. Epub 2014 May 11. PMID 24827808